CLINICAL TRIAL: NCT07040163
Title: Prospective Single-Blinded Randomized Study of Ketamine/Midazolam Deep Sedation vs. Fentanyl/Midazolam Moderate Sedation for Image-Guided Percutaneous Procedures in Interventional Radiology
Brief Title: Evaluation of Ketamine/Midazolam Deep Sedation vs. Fentanyl/Midazolam Moderate Sedation for Image-Guided Percutaneous Procedures in Interventional Radiology
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: CAMC Health System (Other)
Collaborators: Sarah & Pauline Maier Foundation, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 24-1149
Record Dates: First submitted 2025-05-29; First posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Sedation; Interventional Radiology; Biopsy; Drainage Procedure
Keywords: ketamine; interventional radiology; fentanyl; sedation
MeSH Terms: interventions — Ketamine; Fentanyl; Midazolam

STUDY DESIGN:
Intervention Model Description: In this prospective, single-center, single-blind randomized study, all patients 18 years of age and older undergoing image-guided lung and bone biopsy and percutaneous drainage who are eligible for moderate or deep sedation will be recruited. Subjects will be randomized to receive fentanyl/midazolam or ketamine/midazolam using SPSS. Patients will be unaware of which regimen they ultimately receive.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketamine Sedation (Experimental): This arm will utilize a ketamine/midazolam combination sedation for interventional radiology procedures instead of fentanyl/midazolam combination sedation.
  Interventions: Drug: ketamine; Drug: Midazolam
- Fentanyl Sedation (Active Comparator): This arm of the study will receive the traditional fentanyl/midazolam combination sedation for the interventional radiology procedure.
  Interventions: Drug: fentanyl; Drug: Midazolam

INTERVENTIONS:
Drug: ketamine — This is the experimental intervention to be used as an alternative sedation method to the other comparator intervention (fentanyl).
  Arms: Ketamine Sedation
Drug: fentanyl — This is the traditional (comparator) intervention used in interventional radiology procedure sedation.
  Arms: Fentanyl Sedation
Drug: Midazolam — Adjuvant administered in combination with either fentanyl (comparator) or ketamine (experimental).

SUMMARY:
This study aims to reduce pain during interventional radiology (IR) procedures, making the experience better for patients. Typically, doctors use medications like fentanyl and midazolam for sedation. This research will focus on patients undergoing biopsies and drainage procedures, often associated with significant discomfort. Patients will be randomly assigned to receive either fentanyl/midazolam or ketamine/midazolam combinations for sedation. A coordinator will collect information on pain levels and satisfaction, as well as monitor any extra medications needed and side effects. The investigators hope to find that ketamine helps decrease pain and improves satisfaction compared to fentanyl, without increasing complications.

DETAILED DESCRIPTION:
This project will provide the following major innovations:

1. Improve patient experience and satisfaction: Prospective demonstration that ketamine/midazolam results in decreased peri-procedure pain scores and increased satisfaction scores would justify the use of deep sedation in IR and potentially benefit thousands of patients undergoing painful procedures in IR units across the country.
2. Demonstrate the safety and feasibility of ketamine/midazolam sedation administered by IR providers: Showing that performing IR procedures with ketamine/midazolam is as safe or safer than performing the same procedures with fentanyl/midazolam will increase the scope of cases that IR providers can perform without the direct assistance of anesthesia providers and need for recovery in post-anesthesia care units.
3. Provide high level data to justify creation of societal guidelines: One barrier to IR physicians performing deep sedation may be an inability to obtain hospital privileges. Emergency medicine physicians have created societal guidelines to describe the use of deep sedation, enabling successful credentialing. Publishing high quality studies showing safety and efficacy would provide a framework for IR-specific practice guidelines.

The aims of the study are as follows:

Aim 1: Prospectively compare pain and satisfaction scores in patients undergoing IR procedures with either fentanyl/midazolam or ketamine/midazolam. Patients undergoing image-guided biopsy and drainage procedures will be randomized to receive fentanyl/midazolam or ketamine/midazolam. Patients' pain will be rated using the validated 10-point Numeric Rating Scale before, during and after the procedure, and be given questionnaires based on validated anesthesia satisfaction surveys after the procedure to assess their perception of the sedation regimen. Patient groups will be compared in terms of differences on pain scores and the satisfaction survey using two-tailed Mann-Whitney tests.

Aim 2: Prospectively compare the safety of using fentanyl/midazolam or ketamine/midazolam for sedation during IR procedures. Patient groups will be compared in terms of procedure-related adverse events (e.g., hemorrhage, pneumothorax) and sedation-related adverse events (e.g., respiratory compromise) using Fisher's exact tests.

ELIGIBILITY:
Inclusion Criteria:

* Planned to undergo image-guided bone biopsy, lung biopsy, or percutaneous drainage
* Eligible to receive ketamine or fentanyl sedation
* Any sex/gender, any race
* Aged 18-89

Exclusion Criteria:

* Pregnant/lactating
* Incarceration
* Currently taking an opioid agonist/antagonist
* Food consumed in past 6-8 hours
* Allergies to drugs used in the study
* Lacks mental capacity for reporting pain scores
* Hypotension or respiratory failure precluding fentanyl sedation
* Uncontrolled hypertension precluding ketamine sedation
* Condition for which hypertension would be a concern
* Schizophrenia

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Estimated)
Dates: Start 2025-03-07 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Patient's Opinion Survey: Adequacy of Sedation Care | Peri-anesthetic (minimum of 2 hours post-surgery)
  The Adequacy of Sedation Care survey form (a modified version of the Heidelberg peri-anesthetic questionnaire) consists of 18 questions relating to the patient's opinion of the sedation they received. Questions 1-16 are rated on a scale from 1 (Strongly Disagree) to 4 (Strongly Agree). Question 17 asks if the patient would, in the future, have "more sedation," "same sedation," or "less sedation." Question 18 asks the patient to rate their level of pain on a scale from 0 (no pain) to 10 (worst possible pain). It will be administered after the patient has fully recovered from anesthesia, at a minimum of 2 hours post-surgery, well-enough to be discharged from the recovery room.
Numeric Rating Scale (NRS) pain score | Baseline, peri-procedure, peri-anesthetic (minimum 2 hours post-procedure)
  The patient will be asked to assess their pain based on the NRS 11-point pain score system from 0 (no pain) to 10 (worst possible pain) at three different time points: before the procedure (pre-procedure), during the procedure (intra-procedure), and after the procedure (peri-procedure). If the patient does not recall the procedure, it will be marked as a "0" for the intra-procedural portion.

SECONDARY OUTCOMES:
Surgical Procedure and Recovery Time | Start of the procedure, end of the procedure, and when the patient fully recovers from anesthesia well-enough to be discharged from the recovery room. These events (enrollment, procedure, and anesthesia recovery) all occur within the same day.
  The start and end time of the procedure will be recorded, as well as the time it takes for the patient to recover well-enough from anesthesia (minimum of 2 hours post procedure) to be discharged from the recovery room.

CONTACTS AND LOCATIONS:
Overall Officials: Amy R Deipolyi, M.D., Ph.D., Principal Investigator — CAMC Department of Interventional Radiology
Locations (1):
- CAMC Memorial, Charleston, West Virginia, United States

IPD SHARING:
Plan to Share IPD: No
The data obtained from this study relies on patient opinion surveys and pain scales. At this time, individual patient data will not be shared. Data that is relevant to the outcomes of the study, as well as detailed statistical methods, will be included in publications that use the data gathered from this trial.

REFERENCES:
- [Background] Sener S, Eken C, Schultz CH, Serinken M, Ozsarac M. Ketamine with and without midazolam for emergency department sedation in adults: a randomized controlled trial. Ann Emerg Med. 2011 Feb;57(2):109-114.e2. doi: 10.1016/j.annemergmed.2010.09.010. PMID 20970888
- [Background] Radvansky BM, Shah K, Parikh A, Sifonios AN, Le V, Eloy JD. Role of ketamine in acute postoperative pain management: a narrative review. Biomed Res Int. 2015;2015:749837. doi: 10.1155/2015/749837. Epub 2015 Oct 1. PMID 26495312
- [Background] Lemos JN, Lemos LDCN, Solla DJF, Lemos DDCN, Modolo NSP. Patient satisfaction in ambulatory anesthesia assessed by the Heidelberg Peri-anaesthetic Questionnaire: a cross-sectional study. Braz J Anesthesiol. 2023 May-Jun;73(3):258-266. doi: 10.1016/j.bjane.2021.12.003. Epub 2021 Dec 25. PMID 34963617
- [Background] Hawker GA, Mian S, Kendzerska T, French M. Measures of adult pain: Visual Analog Scale for Pain (VAS Pain), Numeric Rating Scale for Pain (NRS Pain), McGill Pain Questionnaire (MPQ), Short-Form McGill Pain Questionnaire (SF-MPQ), Chronic Pain Grade Scale (CPGS), Short Form-36 Bodily Pain Scale (SF-36 BPS), and Measure of Intermittent and Constant Osteoarthritis Pain (ICOAP). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S240-52. doi: 10.1002/acr.20543. No abstract available. PMID 22588748
- [Background] Cashman JN, Ng L. The management of peri- and postprocedural pain in interventional radiology: a narrative review. Pain Manag. 2017 Nov;7(6):523-535. doi: 10.2217/pmt-2017-0024. Epub 2017 Nov 10. PMID 29125398
- [Background] Sutley SH, Kraut RA. A comparison of transcutaneous PO2 in patients sedated with diazepam-fentanyl or midazolam-fentanyl. Anesth Prog. 1989 May-Jun;36(3):93-7. PMID 2638156
- [Background] Boggs SD, Barnett SR, Urman RD. The future of nonoperating room anesthesia in the 21st century: emphasis on quality and safety. Curr Opin Anaesthesiol. 2017 Dec;30(6):644-651. doi: 10.1097/ACO.0000000000000528. PMID 28984638

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-03-07): https://cdn.clinicaltrials.gov/large-docs/63/NCT07040163/Prot_SAP_000.pdf
  • Informed Consent Form (2025-03-07): https://cdn.clinicaltrials.gov/large-docs/63/NCT07040163/ICF_001.pdf